CLINICAL TRIAL: NCT07244575
Title: Association Between Preoperative Metformin Exposure and Postoperative Nausea and Vomiting in Patients Undergoing General Anesthesia: a Prospective Observational Cohort Study
Brief Title: Association Between Preoperative Metformin Exposure and Postoperative Nausea and Vomiting in Patients Undergoing General Anesthesia
Acronym: Met-PONV
Status: Recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yang Zhao, Dr, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: E2025278
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples and urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure group: Patients are already prescribed metformin before surgery
- The non-exposure group: Patients are not prescribed metformin before surgery

SUMMARY:
The aim of this observational study is to investigate the potential effects of metformin on postoperative nausea and vomiting (PONV) in patients undergoing surgery under general anesthesia. The primary research question is:

Does preoperative metformin exposure influence the incidence or severity of PONV in patients undergoing general anesthesia? Patients who are already prescribed metformin as part of their routine medical management will be compared with those not taking metformin. Data on PONV occurrence, severity, and recovery outcomes will be collected through structured postoperative surveys administered after surgery.

DETAILED DESCRIPTION:
This is a prospective observational cohort study involving patients undergoing surgery under general anesthesia with endotracheal intubation at the Sixth Affiliated Hospital of Sun Yat-sen University. A total of 909 participants will be enrolled into either the metformin-exposed group (n=303) or the non-exposed group (n=606) . The primary outcome is the incidence of postoperative nausea and vomiting (PONV) within 0-120 hours after surgery. Secondary outcomes comprise the incidence and severity of PONV during different intervals, use of antiemetics, and quality of recovery (assessed by the QoR-15 score).

ELIGIBILITY:
Inclusion criteria

1. Voluntarily sign the informed consent form;
2. Age ≥ 18 years;
3. Patients who require surgical treatment under endotracheal intubation with general anesthesia as determined by the treating physician.

Exclusion criteria

1. Emergency surgery;
2. Currently taking medications with established antiemetic effects (e.g., corticosteroids, antipsychotics) due to underlying medical conditions;
3. Cognitive impairment or psychiatric disorders that preclude cooperation with questionnaire assessments;
4. Anticipated inability to extubate the tracheal tube postoperatively, which would interfere with outcome assessment;
5. Presence of nausea and/or vomiting prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgery under general anesthesia with tracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 909 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of PONV during 0-120 postoperative hours | During 0-120 hour after surgery
  PONV is defined as the occurrence of any of the following symptoms: nausea, retching, or vomiting

SECONDARY OUTCOMES:
The incidence PONV during 0-24 hour after surgery | During 0-24 hour after surgery
  PONV is defined as the occurrence of any of the following symptoms: nausea, retching, or vomiting
The incidence PONV during 24-120 hour after surgery | During 24-120 hour after surgery
  Trained blinded investigators collected information about PONV recorded by either the participants and their family members or medical staff in the ward every 24 h during the first 120 h after surgery.
The total severity of PONV during 0-120 hour after surgery | During 0-120 hour after surgery
  Assessment was performed using a simplified Postoperative Nausea and Vomiting (PONV) Impact Scale. Nausea severity was scored as follows: 0 (none), 1 (occasional), 2 (frequent), and 3 (continuous). Vomiting or retching was scored based on the number of episodes: 0, 1, 2, or 3 (or ≥3 episodes). The scores for nausea and vomiting/retching were summed to generate a total daily score for each 24-hour postoperative period. A total daily score of ≥5 was defined as clinically significant PONV. The overall PONV severity from 0 to 120 hours postoperatively was calculated as the sum of the daily scores over this period, providing a cumulative measure of symptom burden.
The severity of PONV during 0-24 hour after surgery | During 0-24 hour after surgery
  Assessment was performed using a simplified Postoperative Nausea and Vomiting (PONV) Impact Scale. Nausea severity was scored as follows: 0 (none), 1 (occasional), 2 (frequent), and 3 (continuous). Vomiting or retching was scored based on the number of episodes: 0, 1, 2, or 3 (or ≥3 episodes). The scores for nausea and vomiting/retching were summed to generate a total daily score for each 24-hour postoperative period. A total daily score of ≥5 was defined as clinically significant PONV.
The severity of PONV during 24-120 hour after surgery | During 24-120 hour after surgery
  Assessment was performed using a simplified Postoperative Nausea and Vomiting (PONV) Impact Scale. Nausea severity was scored as follows: 0 (none), 1 (occasional), 2 (frequent), and 3 (continuous). Vomiting or retching was scored based on the number of episodes: 0, 1, 2, or 3 (or ≥3 episodes). The scores for nausea and vomiting/retching were summed to generate a total daily score for each 24-hour postoperative period. A total daily score of ≥5 was defined as clinically significant PONV. The overall PONV severity from 25 to 120 hours postoperatively was calculated as the sum of the daily scores over this period.
Use of antiemetics during 0-24 hours after surgery | During 0-24 hours after surgery
  Use of antiemetics after surgery
Use of antiemetics during 24-120 hours after surgery | During 24-120 hours after surgery
  Use of antiemetics after surgery
Use of antiemetics during 0-120 hours after surgery | During 0-120 hours after surgery
  Use of antiemetics after surgery
Quality of Recovery (QoR-15 score) from 0 to 120 hour after surgery | Evaluated before surgery, at 24-hour, 48-hour, 72-hour, 96-hour, 120-hour after surgery
  The QoR-15 is a 15-item questionnaire instrument designed to evaluate the quality of postoperative recovery in patients. It comprises five sub-scales: pain (2 items), physical comfort (5 items), physical independence (2 items), psychological support (2 items), and emotional state (4 items). Each item is scored from 0 to 10, resulting in a total score ranging from 0 to 150. A higher score indicates a better quality of recovery for the patient.

OTHER OUTCOMES:
Quality of recovery at 30-day after surgery | At 30-day after surgery
  The QoR-15 is a 15-item questionnaire instrument designed to evaluate the quality of postoperative recovery in patients. It comprises five sub-scales: pain (2 items), physical comfort (5 items), physical independence (2 items), psychological support (2 items), and emotional state (4 items). Each item is scored from 0 to 10, resulting in a total score ranging from 0 to 150. A higher score indicates a better quality of recovery for the patient.
Incidence and grade of major postoperative complications | During 30 day after surgery
  Incidence and grade of major postoperative complications
PONV-related factors in the blood or urine. | from preoperative to postoperative
  PONV-related factors in the blood or urine
Overall survival rates | 1-year, 3-year, 5-year after surgery
  The status of live or death, and the death time
Disease-free survival rates at 1-year, 3-year and 5-year, assessed exclusively among patients with cancer. | 1-year, 3-year and 5-year after surgery
  Disease-free survival rates

CONTACTS AND LOCATIONS:
Overall Officials: Yang Zhao, Dr, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available after the manuscript is published.
Access Criteria: The request for the analytic code shall be sent to Prof. Yang Zhao, Email-address: zhaoy47@mail.sysu.edu.cn

REFERENCES:
- [Background] Kincaid JWR, Rimmington D, Tadross JA, Cimino I, Zvetkova I, Kaser A, Richards P, Patel S, O'Rahilly S, Coll AP. The gastrointestinal tract is a major source of the acute metformin-stimulated rise in GDF15. Sci Rep. 2024 Jan 22;14(1):1899. doi: 10.1038/s41598-024-51866-2. PMID 38253650
- [Background] Bootcov MR, Bauskin AR, Valenzuela SM, Moore AG, Bansal M, He XY, Zhang HP, Donnellan M, Mahler S, Pryor K, Walsh BJ, Nicholson RC, Fairlie WD, Por SB, Robbins JM, Breit SN. MIC-1, a novel macrophage inhibitory cytokine, is a divergent member of the TGF-beta superfamily. Proc Natl Acad Sci U S A. 1997 Oct 14;94(21):11514-9. doi: 10.1073/pnas.94.21.11514. PMID 9326641
- [Background] Al-Kuraishy HM, Al-Gareeb AI, Alexiou A, Papadakis M, Nadwa EH, Albogami SM, Alorabi M, Saad HM, Batiha GE. Metformin and growth differentiation factor 15 (GDF15) in type 2 diabetes mellitus: A hidden treasure. J Diabetes. 2022 Dec;14(12):806-814. doi: 10.1111/1753-0407.13334. Epub 2022 Nov 28. PMID 36444166
- [Background] Bu XS, Zhang J, Zuo YX. Validation of the Chinese Version of the Quality of Recovery-15 Score and Its Comparison with the Post-Operative Quality Recovery Scale. Patient. 2016 Jun;9(3):251-9. doi: 10.1007/s40271-015-0148-6. PMID 26518201
- [Background] Myles PS, Wengritzky R. Simplified postoperative nausea and vomiting impact scale for audit and post-discharge review. Br J Anaesth. 2012 Mar;108(3):423-9. doi: 10.1093/bja/aer505. Epub 2012 Jan 29. PMID 22290456
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Sharma N, MacGibbon KW, Brecht-Doscher A, Cortessis VK, Fejzo MS. Prepregnancy metformin use associated with lower risk of severe nausea and vomiting of pregnancy and hyperemesis gravidarum. Am J Obstet Gynecol. 2025 Dec;233(6):649.e1-649.e14. doi: 10.1016/j.ajog.2025.06.055. Epub 2025 Jun 28. PMID 40588059
- [Background] Sillis L, Heinonen EW, Ceulemans M, Johnson D, Luo Y, Chambers CD. Metformin for the Prevention of Hyperemesis Gravidarum: An Observational Cohort Study. BJOG. 2025 Nov;132(12):1772-1778. doi: 10.1111/1471-0528.18238. Epub 2025 May 29. PMID 40443168
- [Background] Day EA, Ford RJ, Smith BK, Mohammadi-Shemirani P, Morrow MR, Gutgesell RM, Lu R, Raphenya AR, Kabiri M, McArthur AG, McInnes N, Hess S, Pare G, Gerstein HC, Steinberg GR. Metformin-induced increases in GDF15 are important for suppressing appetite and promoting weight loss. Nat Metab. 2019 Dec;1(12):1202-1208. doi: 10.1038/s42255-019-0146-4. Epub 2019 Dec 9. PMID 32694673
- [Background] Mai Y, Zhang S, Huang Q, Liang C, Shi J, Zheng J, Lv K, Liu H, Yang X, Zhao Y. Association between plasma growth differentiation factor-15 and postoperative nausea and vomiting incidence and severity: a secondary analysis of a randomised trial. Br J Anaesth. 2025 Aug;135(2):459-468. doi: 10.1016/j.bja.2025.05.001. Epub 2025 May 29. PMID 40441987
- [Background] Hsu JY, Crawley S, Chen M, Ayupova DA, Lindhout DA, Higbee J, Kutach A, Joo W, Gao Z, Fu D, To C, Mondal K, Li B, Kekatpure A, Wang M, Laird T, Horner G, Chan J, McEntee M, Lopez M, Lakshminarasimhan D, White A, Wang SP, Yao J, Yie J, Matern H, Solloway M, Haldankar R, Parsons T, Tang J, Shen WD, Alice Chen Y, Tian H, Allan BB. Non-homeostatic body weight regulation through a brainstem-restricted receptor for GDF15. Nature. 2017 Oct 12;550(7675):255-259. doi: 10.1038/nature24042. Epub 2017 Sep 27. PMID 28953886
- [Background] Cheng W, Gordian D, Ludwig MQ, Pers TH, Seeley RJ, Myers MG Jr. Hindbrain circuits in the control of eating behaviour and energy balance. Nat Metab. 2022 Jul;4(7):826-835. doi: 10.1038/s42255-022-00606-9. Epub 2022 Jul 25. PMID 35879458
- [Background] Borner T, Tinsley IC, Milliken BT, Doebley SA, Najjar NR, Kerwood DJ, De Jonghe BC, Hayes MR, Doyle RP. Creation of a Peptide Antagonist of the GFRAL-RET Receptor Complex for the Treatment of GDF15-Induced Malaise. J Med Chem. 2023 Aug 24;66(16):11237-11249. doi: 10.1021/acs.jmedchem.3c00667. Epub 2023 Jul 28. PMID 37506293
- [Background] Liu ZY, Yang XY, Lv C, Ye L, Chen JJ, Chen XY, Wang SP, Wu L, Zhang WQ, Lu M, Guo XW. Effect of High Maintenance Dose Versus Low Dose of Remifentanil on Incidence of Postoperative Nausea and Vomiting (PONV) in Patients Under Gynecological Laparoscopic Procedure: A Pilot Study. Drug Des Devel Ther. 2025 Jun 7;19:4885-4894. doi: 10.2147/DDDT.S518291. eCollection 2025. PMID 40502550
- [Background] Zhang Q, Ye X, Shi S, Zhou S, Ma D, Ouyang W, Tong J, Le Y. Pyridoxine Prevents Postoperative Nausea and Vomiting in Gynecologic Laparoscopic Surgery: A Double-blind Randomized Controlled Trial. Anesthesiology. 2025 Apr 1;142(4):655-665. doi: 10.1097/ALN.0000000000005354. Epub 2024 Dec 27. PMID 39729294